CLINICAL TRIAL: NCT03090022
Title: Prophylactic Mesh Implantation in Patients Undergoing Requiring Emergency Laparatomy for the Prevention of Incisional Hernia:A Randomized Controlled Trial
Brief Title: Hernia-Prophylaxis in Acute Care Surgery H-PACS
Acronym: H-PACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2016-02212
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia | interventions — strattice

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesh implantation (Active Comparator): Prior to closure of the abdominal wall a mesh will be implanted in a standardized fashion
  Interventions: Procedure: Strattice
- Single running suture of abdominal fascia (Active Comparator): The closure of the abdominal wall a Standard technique will be applied using a running suture
  Interventions: Procedure: Single running suture of abdominal fascia

INTERVENTIONS:
Procedure: Strattice — Intra-abdominally Fixation
  Other Names: Acellular porcine dermal mesh
  Arms: Mesh implantation
Procedure: Single running suture of abdominal fascia — Intra-abdominal suture
  Arms: Single running suture of abdominal fascia

SUMMARY:
Incisional hernia is a common complication in visceral surgery and varies between 11 and 26% in the general surgical population. Patients requiring emergency laparotomy are at high risk for the development of incisional hernia and fascial dehiscence. Among this population the incidence of incisional hernia in patients undergoing emergency surgery varies between 33-54%. Incisional hernias are associated with a high morbidity rate, such as intestinal incarceration, chronic discomfort, pain, and reoperation and typically require implantation of a synthetic mesh in a later second operation. Fascial dehiscence represents an acute form of dehiscence and has been observed in up to 24.1% and is associated with a mortality rate up to 44%.

The gold standard for abdominal wall closure during elective and emergency operations is a running slowly absorbable suture. In the elective situation it has been shown that prophylactic mesh implantation in high risk patients reduced the incidence of incisional hernia significantly.

The investigators and others have shown that mesh implantation in patients undergoing emergency laparotomy or in contaminated abdominal cavities are safe .

With a randomized controlled trial the investigators now aim to compare the incidence of incisional hernia after prophylactic mesh implantation versus standard of care in patients requiring emergency laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing emergency midline laparatomy
* Emergency laparoscopy with expected conversion to midline laparatomy
* Written informed consent

Exclusion Criteria:

* ASA ≥5
* Septic shock
* Pregnant women
* Prior mesh Implantation
* Known sensitivity for porcine material or Polysorbate 20

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Number of incidence of death | up to 18 months
  follow-up
Number of patients with hernia free survival | up to 18 months
  follow-up

SECONDARY OUTCOMES:
Number of patients with postoperative fascial dehiscence | 30 days
  follow-up
Number of postoperative mortality | 90 days
  survival
Number of surgical site infections postoperative | 30 days
  follow-up
Number of postoperative intestinal fistulas | 30 days
  follow-up
Number of small bowel obstructions | 18 months
  follow-up
Number of patients with postoperative pain | 18 months
  follow-up
Number of postoperative mesh infections | 18 months
  follow-up
Number of postoperative mesh explantations | 18 months
  follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Guido Beldi, Prof. Dr., Principal Investigator — Inselspital Berne
Locations (1):
- Dep. of Visceral and transplant surgery, Berne University Hospital, Bern, Switzerland